CLINICAL TRIAL: NCT04077411
Title: Approaches and Decisions for Acute Pediatric TBI (ADAPT) Trial
Brief Title: Approaches and Decisions for Acute Pediatric TBI Trial
Acronym: ADAPT
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Stephen Wisniewski, Professor, University of Pittsburgh
Other Study IDs: PRO13020047; U01NS081041 (NIH)
Record Dates: First submitted 2019-08-29; First posted 2019-09-04 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-03

CONDITIONS: Severe Traumatic Brain Injury
Keywords: Severe Traumatic Brain Injury; TBI; Intracranial hypertension; Cerebrospinal fluid; Hypersmolar therapies; Prophylactic hyperventilation; Metabolism; Neuropsychology
MeSH Terms: conditions — Brain Injuries, Traumatic; Intracranial Hypertension | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with severe TBI: Children with severe Traumatic Brain Injury
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — This is an observational study with no interventions.

SUMMARY:
Approaches and Decisions in Acute Pediatric TBI Trial (ADAPT) is an international research study designed to evaluate the impact of interventions on the outcomes of children with severe traumatic brain injury.

Pediatric traumatic brain injury (TBI) is the leading killer of children, resulting in more than 7000 deaths and $2 billion in acute care costs each year. Despite this large burden of disease, advances in the field have been limited due to weak evidenced-based guidelines and the limitations of randomized, controlled trials (RCTs) to demonstrate efficacy of single treatment strategies due to wide treatment variability. ADAPT is a practical study design in a novel approach - an observational cohort study designed to evaluate the association of 6 aspects of pediatric TBI care with outcomes using statistical modeling to correct for confounding variables. Completion of this study will provide compelling evidence to change clinical practices, provide evidence for new Level II recommendations for future guidelines and lead to improved research protocols that would limit variability in TBI treatments - helping children immediately through better clinical practices and ultimately through more effective investigation.

DETAILED DESCRIPTION:
Traumatic brain injury (TBI) is the leading cause of death in children in the US. According to the CDC, 7440 children died of TBI in 2005, but this likely underestimates the full burden of the disease. Based on the current best estimates for severe pediatric TBI (20% mortality, 50.6% unfavorable 6 mo outcome, mean age 9 y), each year 37,200 children suffer a severe TBI with up to 1.3 million life-years potentially adversely affected.

Incremental improvement in outcomes could make enormous differences for the health of children, but such advances have remained elusive. Dozens of injury mechanisms have been identified after experimental TBI, yet no mitigating treatments have been translated into clinical practice. Randomized controlled trials (RCTs) of therapies, from steroids to novel pharmaceutical agents to hypothermia, have failed for adult and pediatric TBI victims. Single-center experiences have contributed to understanding, yet these largely remain insufficiently powerful to change practice. Recently, evidenced-based guidelines for 15 aspects of pediatric TBI were published that provide no level I and only 4 Level II recommendations - with such recommendations indicating therapies that "must be done" or "should be considered" based on the literature, respectively. Disappointingly, 3 of these recommendations advised against specific interventions (hypothermia, steroids and immune-enhanced diets) - emphasizing the uncertainty of the effectiveness of many commonly used therapies that leads to wide variations in clinical practice. Unsurprisingly, significant variations of clinical outcomes and basic treatment strategies for TBI have been observed. The IMPACT study merged data from over 9000 adults with TBI from 11 trials and demonstrated significant variations in outcomes from clinical sites. Similar variations in outcomes in children with TBI can be found using various administrative databases, with mortality rates varying between 12.2% - 34.4% in 11 US states. There are also variations in strategies within an international consortium and a recently completed RCT - with marked variations in strategies for first-line intracranial hypertension treatments, prevention of common secondary insults and metabolic support after pediatric TBI.

The paucity of data to create robust guidelines, the failure of RCTs that tested a wide-variety of putative mechanisms and variations in outcomes and in clinical practices argues that the current understanding of contemporary therapies is inadequate. Because neither retrospective analyses from available databases nor self-reported variations in practices can determine optimal therapeutic strategies for these contemporaneous strategies, a new approach is urgently needed.

ADAPT is a large, prospective, observational cohort study using an international consortium including sites from the US, EU and UK. Children with severe TBI [Glasgow coma scale (GCS) score ≤ 8 with intracranial pressure (ICP) monitoring, n = 1000, >32 sites] will be studied. The local standard of care at each site will be used and extensive data collection over the first 7 days after TBI will be performed to interrogate the effectiveness of strategies for intracranial hypertension, mitigation of specific secondary insults and metabolism.

Several statistical approaches, often used in comparative effectiveness research (CER) to control for measured confounding effects, will test the following aims:

Specific Aim 1: Compare the effectiveness of first-line intracranial hypertension strategies on outcome. Intracranial hypertension management is a mainstay of TBI care yet evidence for utilization the first-line therapies of cerebrospinal fluid (CSF) diversion and use of hyperosmolar solutions, is incomplete.

Aim 1a: Determine the effect of CSF diversion strategies (continuous drainage, intermittent drainage and none) on outcome. Aim 1b: Determine the effect of hyperosmolar therapies (hypertonic saline, mannitol) on outcome.

Specific Aim 2: Compare the effectiveness of strategies that mitigate specific secondary insults on outcome. Prophylactic hyperventilation (HV) and hypoxia may worsen outcome after TBI but have been inadequately studied.

Aim 2a: Determine the effect of prophylactic HV (CO2 < 30 mm Hg) on outcome.

Aim 2b: Determine the effect of hypoxia detection with brain tissue oxygen monitoring (PbO2) on outcome.

ELIGIBILITY:
Inclusion Criteria:

* Admission to a study site for treatment of severe traumatic brain injury
* ICP monitor placed as part of the child's standard care
* Glasgow Coma Scale (GCS) ≤ 8 after resuscitation
* Age 0 - 18 y

Exclusion Criteria:

* 1. ICP Monitor placed at another hospital
* 2. Diagnosis of pregnancy in clinical subject

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with severe traumatic brain injury (TBI)
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2014-02-20 (Actual); Primary Completion 2016-09-26 (Actual); Study Completion 2018-08-28 (Actual)

PRIMARY OUTCOMES:
Glasgow Outcome Score - Extended Pediatrics | 6 months
  Physician-rated assessment of functional outcome. Problems in functioning should have deteriorated from premorbid level. The categories are:
  8 - Death 7 - Vegetative State (VS) 6 - Lower Severe Disability (Lower SD) 5 - Upper Severe Disability (Upper SD) 4 - Lower Moderate Disability (Lower MD) 3 - Upper Moderate Disability (Upper MD) 2 - Lower Good Recovery (Lower GR)
  1 - Upper Good Recovery (Upper GR)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Bell, MD, Principal Investigator — University of Pittsburgh Medical Center; Stephen R Wisniewski, PhD, Principal Investigator — University of Pittsburgh
Locations (48):
- United States (30):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - University of California, San Diego / Rady's Children's Hospital, La Jolla, California
  - Children's Hospital of Los Angeles, Los Angeles, California
  - UCLA Mattel Children's Hospital, Los Angeles, California
  - UC Davis Medical Center, West Sacramento, California
  - Children's Hospital Colorado, Denver, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Miami Children's Hospital, Miami, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - University of Iowa Children's Hospita, Iowa City, Iowa
  - John Hopkins Children's Center of Baltimore, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Children's Hospital / Harvard University, Boston, Massachusetts
  - Wayne State University in Detroit / Children's Hospital of Michigan, Detroit, Michigan
  - Washington University - St. Louis, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Carolinas Medical Center Levine Children's Hospital, Charlotte, North Carolina
  - University of Cincinnati / Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Penn State University - Hershey, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - University of Tennessee / Le Bonheur Children's Hospita, Memphis, Tennessee
  - UT Southwestern / Children's Medical Center at Dallas, Dallas, Texas
  - Texas Children's Hospital (Baylor College of Medicine), Houston, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Children's Hospital of Richmond at VCU, Richmond, Virginia
  - University of Washington - Seattle, Seattle, Washington
  - University of Wisconsin - Madison, Madison, Wisconsin
- Australia (3):
  - Children's Health Queensland Hospital and Health Service, Brisbane
  - Royal Children's Hospital, Melbourne
  - Princess Margaret Hospital, Perth
- All India Institute of Medical Sciences, New Delhi, India
- Erasmus Medical Center Children's Hospital, Rotterdam, Netherlands
- Starship Children's Hospital, Auckland, New Zealand
- University of Cape Town, Cape Town, South Africa
- Hospital Vall d'Hebron, Barcelona, Spain
- United Kingdom (10):
  - Birmingham Children's Hospita, Birmingham
  - University Hospitals Bristol, Bristol
  - Addenbrookes Hospital, Cambridge
  - Leeds Teaching Hospital, Leeds
  - Alder Hey Children's, Liverpool
  - King's College Hospital, London
  - Great Ormond Street, London
  - Newcastle upon Tyne Hospital, Newcastle upon Tyne
  - University Hospital Southampton, Southampton
  - Royal Manchester Children's Hospital, Victoria

IPD SHARING:
Plan to Share IPD: Yes
Study data will be released to the general public through FITBIR. ADAPT will adhere to all FITBIR policies and procedures.
Supporting Information: Study Protocol, ICF
Time Frame: One year after publication of main results paper.
Access Criteria: Investigators requesting and receiving FITBIR data are expected to:
  * Submit a Data Access Request;
  * Protect data confidentiality;
  * Ensure that data security measures are in place;
  * Notify the Data Access and Quality Committee of policy violations;
  * Submit annual progress reports detailing significant research findings; and
  * Include acknowledgements of the FITBIR Informatics System in all publications and presentations.

REFERENCES:
- [Background] Sarnaik A, Ferguson NM, O'Meara AMI, Agrawal S, Deep A, Buttram S, Bell MJ, Wisniewski SR, Luther JF, Hartman AL, Vavilala MS; Investigators of the ADAPT Trial. Age and Mortality in Pediatric Severe Traumatic Brain Injury: Results from an International Study. Neurocrit Care. 2018 Jun;28(3):302-313. doi: 10.1007/s12028-017-0480-x. PMID 29476389
- [Background] Bell MJ, Adelson PD, Wisniewski SR; Investigators of the ADAPT Study,. Challenges and opportunities for pediatric severe TBI-review of the evidence and exploring a way forward. Childs Nerv Syst. 2017 Oct;33(10):1663-1667. doi: 10.1007/s00381-017-3530-y. Epub 2017 Sep 6. PMID 29149394
- [Background] Miller Ferguson N, Sarnaik A, Miles D, Shafi N, Peters MJ, Truemper E, Vavilala MS, Bell MJ, Wisniewski SR, Luther JF, Hartman AL, Kochanek PM; Investigators of the Approaches and Decisions in Acute Pediatric Traumatic Brain Injury (ADAPT) Trial. Abusive Head Trauma and Mortality-An Analysis From an International Comparative Effectiveness Study of Children With Severe Traumatic Brain Injury. Crit Care Med. 2017 Aug;45(8):1398-1407. doi: 10.1097/CCM.0000000000002378. PMID 28430697
- [Background] Larsen GY, Schober M, Fabio A, Wisniewski SR, Grant MJ, Shafi N, Bennett TD, Hirtz D, Bell MJ. Structure, Process, and Culture Differences of Pediatric Trauma Centers Participating in an International Comparative Effectiveness Study of Children with Severe Traumatic Brain Injury. Neurocrit Care. 2016 Jun;24(3):353-60. doi: 10.1007/s12028-015-0218-6. PMID 26627225
- [Derived] Ahmed N, Russo L, Kuo YH. Levetiracetam or Phenytoin as Prophylaxis for Status Epilepticus: Secondary Analysis of the "Approaches and Decisions in Acute Pediatric Traumatic Brain Injury Trial" (ADAPT) Dataset, 2014-2017. Pediatr Crit Care Med. 2024 Aug 1;25(8):710-719. doi: 10.1097/PCC.0000000000003526. Epub 2024 May 8. PMID 38717237
- [Derived] Surtees TL, Kumar I, Garton HJL, Rivas-Rodriguez F, Parmar H, McCaffery H, Riebe-Rodgers J, Shellhaas RA. Levetiracetam Prophylaxis for Children Admitted With Traumatic Brain Injury. Pediatr Neurol. 2022 Jan;126:114-119. doi: 10.1016/j.pediatrneurol.2021.10.009. Epub 2021 Oct 19. PMID 34839268